CLINICAL TRIAL: NCT02652663
Title: Liver MRI for Colorectal Cancer Liver Metastasis: Comparative Effectiveness Research for the Choice of Contrast Agents
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-1045
Record Dates: First submitted 2016-01-06; First posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; liver; MRI; contrast; gadoxetic acid
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ECA-MRI group: ECA-MRI group (patients who underwent conventional MRI using extracellular contrast agent [ECA])
- Gd-EOB-MRI group: Gd-EOB-MRI group (patients who underwent gadoxetic acid-enhanced MRI)

SUMMARY:
Magnetic resonance imaging (MRI) has been widely used for problem-solving tool in the evaluation of hepatic lesions, and it has been shown to have better sensitivity than CT for detection of colorectal liver metastases, especially for lesions which are smaller than 1 cm. After introduction of a liver-specific hepatobiliary MR contrast agent, gadoxetic acid, gadoxetic acid-enhanced MRI (Gd-EOB-MRI) has been increasingly used for evaluation of liver lesion including CRLM. However, compared to conventional MRI with extracellular contrast agent (ECA-MRI), Gd-EOB-MRI has different pharmacodynamic characteristics, and is more expensive due to higher cost of gadoxetic acid and needs longer scan time to obtain hepatobiliary phase which is generally acquired 15 to 20 minutes after contrast injection. The purpose of this study was to compare the clinical outcome and diagnostic performance of Gd-EOB-MRI and ECA-MRI for evaluation of focal hepatic lesion in newly diagnosed colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. patients with surgically proven colorectal adenocarcinoma
2. patients who underwent abdominopelvic CT and liver MRI for initial staging before any treatment
3. no past or concurrent malignancy other than colorectal adenocarcinoma.

Exclusion Criteria:

1. precontrast abdominopelvic CT
2. precontrast liver MRI
3. liver MRI using contrast other than extracellular agent or gadoxetic acid
4. the interval between CT and liver MRI was longer than 4 weeks
5. patients who had suspected multiple hepatic metastases (> 10) on CT
6. distant metastasis other than liver and
7. unavailable reference standard of their hepatic lesions with no pathologic confirmation or follow up imaging.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed colorectal cancer between January 2005 and December 2010
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | up to 120 months
  From date of curative hepatic surgery until the date of first documented tumor recurrence or date of death from disease-related cause

IPD SHARING:
Plan to Share IPD: No
no plant to shae data